CLINICAL TRIAL: NCT05727449
Title: Comparison of The Effects of General and Spinal Anesthesia for Cesarean Delivery on Maternal and Fetal Outcomes: A Retrospective Analysis of Data in a Third Level Hospital
Brief Title: General or Spinal Anesthesia for Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Medical Doctor, Istanbul Medeniyet University
Other Study IDs: IstanbulMU Cesarean Delivery
Record Dates: First submitted 2023-01-22; First posted 2023-02-14 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Anesthesia for Cesarean Delivery
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia for Cesarean Delivery
  Interventions: Procedure: General Anesthesia
- Spinal Anesthesia for Cesarean Delivery
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — General Anesthesia was intruduced for Cesarean Delivery
  Groups: General Anesthesia for Cesarean Delivery
Procedure: Spinal Anesthesia — Spinal Anesthesia was intraduced for Cesarean Delivery
  Groups: Spinal Anesthesia for Cesarean Delivery

SUMMARY:
During the cesarean deliveries, one of the anesthesia techniques, regional anesthesia or general anesthesia (GA) is prefered. Spinal anesthesia (SA) is preferred among the regional anesthesia methods because the onset of anesthesia is faster and muscle relaxation is more suitable for cesarean section anesthesia. Although both methods have advantages and disadvantages, the anesthesia method to be chosen may vary depending on the condition of the mother and fetus.

The goal of this retrospective clinical trial is to compare general and spinal anesthesia in cesarean deliveries. The main questions it aims to answer are:

* Are the anesthesia techniques effect maternal outcome?
* Are the anesthesia techniques effect fetal outcome?

ELIGIBILITY:
Inclusion Criteria:

The pregnant women who delivered with cesarean section

Exclusion Criteria:

* The pregnant women who delivered with spontan vaginal delivery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The pregnant women and their babies in 01.01.2019 - 31.12.2019.
Sampling Method: Probability Sample
Enrollment: 862 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Apgar 1st minute score | 1st minute after birth
  The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health
Apgar 5th minute score | 5th minute after birth
  The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health
Umbilical Cord Blood pH | at the time of birth
  pH values from umblical cord blood sampling
Umbilical Cord Blood PCO2 | at the time of birth
  mmHg
Umbilical Cord Blood HCO3 | at the time of birth
  mEq/L
Umbilical Cord Blood Lactate | at the time of birth
  mmol/L
Umbilical Cord Blood Base Excess | at the time of birth
  mEq/L
need for neonatal intensive care | up to 24 hours
  need for neonatal intensive care
need for maternal intensive care | up to 24 hours
  need for maternal intensive care

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No